CLINICAL TRIAL: NCT03455270
Title: A Phase 1, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of Ascending Doses of G1T48 Alone and in Combination With Palbociclib in Women With Estrogen Receptor-Positive, HER2-Negative Advanced Breast Cancer
Brief Title: G1T48, an Oral SERD, Alone and in Combination With Palbociclib in ER-Positive, HER2-Negative Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: G1T48-01; 2017-004502-17 (EudraCT Number)
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Carcinoma, Ductal, Breast; Breast Cancer Female; Breast Neoplasm; Breast Cancer; Metastatic Breast Cancer; Advanced Breast Cancer; Stage IV Breast Cancer
Keywords: Breast Cancer; Oral SERD; SERD; HER2-Negative; ER-Positive; ER+; HER2-; HER2 -ve; ER +ve; CDK 4/6 Inhibitor; Rintodestrant; G1T48
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose Escalation (G1T48) (Experimental): Patients in Part 1 will receive a single oral dose of G1T48 on Cycle 1 Day -3 and will begin once-daily dosing on Cycle 1 Day 1.
  The initial dose cohort shall receive an identified starting dose and subsequent cohorts shall receive higher doses based on the safety and PK data obtained from the previous dose levels.
  Interventions: Drug: G1T48
- Part 1: Food Effect Cohort (G1T48) (Experimental): In Part 1, additional G1T48 cohort(s) of 8 patients may be enrolled to assess the effect of different fat content meals (eg, high fat, moderate fat, or low-fat) on the rate and extent of the absorption of G1T48.
  Patients will receive a single oral dose of G1T48 on Cycle 1 Day -10 and on Cycle 1 Day -3. Patients will begin G1T48 once-daily dosing on Cycle 1 Day 1.
  Interventions: Drug: G1T48
- Part 2: Monotherapy Dose Expansion (G1T48) (Experimental): Patients in Part 2 will receive G1T48 once-daily at the dose determined in Part 1.
  Interventions: Drug: G1T48
- Part 3: Combination Dose Expansion (G1T48+palbociclib) (Experimental): Patients in Part 3 will receive G1T48 once-daily at the dose determined in Part 2 in combination with palbociclib once-daily on Days 1 to 21 of each 28-day cycle.
  Interventions: Drug: G1T48; Drug: Palbociclib

INTERVENTIONS:
Drug: G1T48 — oral SERD
  Other Names: Rintodestrant
Drug: Palbociclib — CDK 4/6 Inhibitor
  Other Names: Ibrance
  Arms: Part 3: Combination Dose Expansion (G1T48+palbociclib)

SUMMARY:
This is a study to investigate the potential clinical benefit of G1T48 as an oral selective estrogen receptor degrader (SERD) alone and in combination with palbociclib, a cyclin dependent kinase 4/6 (CDK 4/6) inhibitor, in patients with estrogen receptor-positive, HER2-negative metastatic breast cancer.

The study is an open-label design, consisting of 3 parts: dose-finding portion including food effect (Part 1), G1T48 monotherapy expansion portion (Part 2), and G1T48 in combination with palbociclib expansion portion (Part 3). All parts include 3 study phases: Screening Phase, Treatment Phase, and Survival Follow-up Phase. The Treatment Phase begins on the day of first dose with study treatment and completes at the Post-Treatment Visit. Approximately, 184 patients may be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* For Part 1, postmenopausal women only
* For Parts 2 and 3, any menopausal status
* Confirmed diagnosis of ER-positive, HER2-negative advanced breast cancer, not amenable to curative therapy
* For Part 1, prior treatment with less than 4 prior lines of chemotherapy
* For Part 2, prior treatment with less than 2 prior line of chemotherapy
* For Part 3, prior treatment with no more than 1 prior line of chemotherapy
* For Parts 1 and 2, prior treatment with less than 4 prior endocrine therapies for metastatic breast cancer
* For Part 3, prior treatment with no more than 1 prior line of endocrine therapies for metastatic breast cancer
* For Parts 1 and 2, patients must satisfy 1 of the following criteria for prior therapy:

  * Progressed during treatment or within 12 months of completion of adjuvant therapy with an aromatase inhibitor
  * Progressed after the end of prior aromatase inhibitor therapy for advanced/metastatic breast cancer
* For Part 3, patients must satisfy 1 of the following criteria for prior therapy:

  * Received ≥ 24 months of endocrine therapy in the adjuvant setting prior to recurrence or progression
  * Received ≥ 6 months of endocrine therapy in the advanced/metastatic setting prior to progression
* For Part 1, evaluable or measurable disease
* For Parts 2 and 3, evaluable (approximately 25%) or measurable disease (approximately 75%) as defined by RECIST, Version 1.1 including bone-only disease
* ECOG performance status 0 to 1
* Adequate organ function

Exclusion Criteria:

* For Part 3, prior treatment with CDK4/6 inhibitor, investigational oral SERDs or SERCAs in any setting
* Active uncontrolled/symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease
* Anticancer therapy within 14 days of first G1T48 dose or within 28 days for antibody-based therapy
* Concurrent radiotherapy, radiotherapy within 14 days of first G1T48 dose, previous radiotherapy to the target lesion sites, or prior radiotherapy to > 25% of bone marrow
* Prior hematopoietic stem cell or bone marrow transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 107 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Cycle 1 Day -3 to Cycle 1 Day 28
Recommended Phase 2 dose | 12 months
  G1T48 alone and in combination with palbociclib; progression-free survival (PFS)
Number of Treatment Related Adverse Event, including Abnormal Laboratory Events | 21 months
  All AEs, including clinical laboratory, vitals signs, physical examinations and ECGs will be analyzed in all patients receiving study drug(s) from the signing of the informed consent until 30 days after the last dose of study medication(s).

SECONDARY OUTCOMES:
Tumor response based on RECIST, Version 1.1 | 21 months
  G1T48 alone and in combination with palbociclib;
Effect of food on bioavailability of G1T48 | Part 1, Cycle 1 Day -10 to Cycle 1 Day 1.
Pharmacokinetics of G1T48 and metabolites: Maximum Plasma Concentration (Cmax) | Part 1, Cycle 1 Day -3 to Cycle 2 Day 1. Part 2, Cycle 2 Day 1 to Cycle 3 Day 1. Part 3, Cycle 2 Day 1 to Cycle 3 Day 1.
Pharmacokinetics of G1T48 and metabolites: Area under Curve - plasma concentration (AUC) | Part 1, Cycle 1 Day -3 to Cycle 2 Day 1. Part 2, Cycle 2 Day 1 to Cycle 3 Day 1. Part 3, Cycle 2 Day 1 to Cycle 3 Day 1.
Pharmacokinetics of G1T48 and metabolites: Plasma: terminal half life (T1/2) | Part 1, Cycle 1 Day -3 to Cycle 2 Day 1. Part 2, Cycle 2 Day 1 to Cycle 3 Day 1. Part 3, Cycle 2 Day 1 to Cycle 3 Day 1.
Pharmacokinetics of G1T48 and metabolites: Plasma - Volume of distribution | Part 1, Cycle 1 Day -3 to Cycle 2 Day 1. Part 2, Cycle 2 Day 1 to Cycle 3 Day 1. Part 3, Cycle 2 Day 1 to Cycle 3 Day 1.
Pharmacokinetics of palbociclib: Plasma - Trough concentration | Part 3, Cycle 2 Day 1 to Cycle 3 Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Contact, Study Director — G1 Therapeutics, Inc.
Locations (15):
- United States (6):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Stanford Women Cancer Center, Stanford, California
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - UZ Leuven, Leuven
- MHAT for Womens Health - Nadezhda OOD, Sofia, Bulgaria
- ARENSIA Exploratory Medicine LLC, Tbilisi, Georgia
- ARENSIA Exploratory Medicine Phase I Unit, The Institute of Oncology, Chisinau, Moldova
- Netherlands (3):
  - VU University Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
- Spizhenko Clinic, Kiev, Ukraine